CLINICAL TRIAL: NCT02718261
Title: Sup-Icu RENal (SIREN) - a Sub-analysis of the Prospective SUP (Stress Ulcer Prophylaxis)-ICU Trial on the Risk of GI- Bleeding in ICU Patients Receiving Renal Replacement Therapy
Brief Title: Sup-Icu RENal (SIREN)
Acronym: SIREN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jörg Schefold, SIREN principle investigator, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SIREN
Record Dates: First submitted 2016-03-14; First posted 2016-03-24 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Critical Illness; Acute Kidney Injury; End-stage Renal Disease; Renal Replacement Therapy; Proton Pump Inhibitor
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Kidney Failure, Chronic | interventions — Pantoprazole; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Verum (pantoprazole) (Experimental)
  Interventions: Drug: Pantoprazole
- Placebo (Placebo Comparator): 0.9% saline
  Interventions: Drug: Saline 0.9% (matching placebo)

INTERVENTIONS:
Drug: Pantoprazole
  Arms: Verum (pantoprazole)
Drug: Saline 0.9% (matching placebo)
  Arms: Placebo

SUMMARY:
Data show that episodes of bleeding may often be observed in critically ill patients with dialysis-dependent acute renal failure (ARF) on renal replacement therapy (RRT). From a clinical perspective, patients with dialysis-dependent ARF and end-stage renal disease (ESRD) may be considered a high risk population in regard to e.g. development of gastrointestinal (GI-) bleeding.

In the current prospective subanalysis "SIREN" of the randomized placebo-controlled clinical trial "SUP-ICU" (NCT02467621), the investigators seek to elucidate whether the subpopulation of critically ill patients with acute kidney injury requiring renal replacement therapy (RRT) benefit from prophylactic treatment with a proton-pump-inhibitor such as pantoprazole.

ELIGIBILITY:
Inclusion Criteria:

* please refer to SUP-ICU (NCT02467621) trial

Exclusion Criteria:

* please refer to SUP-ICU (NCT02467621) trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3350 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with clinically important GI bleeding | 90 days or length of ICU stay, as applicable

SECONDARY OUTCOMES:
Proportion of patients with one or more of the following adverse events: clinically important GI bleeding, pneumonia, C. difficile infection, or acute myocardial ischemia in the ICU | 90 days or length of ICU stay, as applicable
Proportion of patients with serious adverse reactions | 90 days or length of ICU stay, as applicable
Proportion of patients with one or more infectious adverse events (pneumonia or CDI) in the ICU | 90 days or length of ICU stay, as applicable
Days alive without use of mechanical ventilation, renal replacement therapy, or circulatory support in the 90-day period | 90 days or length of ICU stay, as applicable
90-day and 1-year (365 days) mortality post-randomization | 90 days/365 days or length of ICU stay, as applicable
Proportion of patients receiving treatment (interventions) to stop GI-bleeding (i.e. endoscopy/ open or laparoscopic surgery/ coiling). | 90 days or length of ICU stay, as applicable
Number of units of packed red blood cells (RBCs) transfused. | 90 days or length of ICU stay, as applicable
90-day/360-day/ ICU mortality rate in "RRT group" vs. "ESRD group" vs. "RRT at any time on the ICU" vs. "control group" incl. analysis of verum/ placebo subgroups. | 90 day, 360 days, or length of ICU stay, as applicable

CONTACTS AND LOCATIONS:
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- Dept. of Intensive Care Medicine, University of Bern,, Bern, Switzerland

REFERENCES:
- [Derived] Schefold JC, Krag M, Marker S, Perner A, Wetterslev J, Wise MP, Borthwick M, Bendel S, Keus F, Guttormsen AB, Lange T, Moller MH; the SUP-ICU investigators. Outcomes of Prophylactic Pantoprazole in Adult Intensive Care Unit Patients Receiving Dialysis: Results of a Randomized Trial. Am J Nephrol. 2019;50(4):312-319. doi: 10.1159/000502732. Epub 2019 Sep 3. PMID 31480045
- [Derived] Schefold JC, Perner A, Lange T, Wetterslev J, Wise MP, Borthwick M, Bendel S, Keus F, Guttormsen AB, Marker S, Krag M, Moller MH; SUP-ICU investigators. Effects of stress ulcer prophylaxis in adult ICU patients receiving renal replacement therapy (Sup-Icu RENal, SIREN): Study protocol for a pre-planned observational study. Trials. 2018 Jan 10;19(1):26. doi: 10.1186/s13063-017-2408-3. PMID 29321041
- See also: Homepage SUP-ICU RCT — http://www.sup-icu.com
- Available data/document: Study Protocol: NCT02467621 — https://clinicaltrials.gov/ct2/show/NCT02467621?term=SUP-ICU&rank=1 — SUP-ICU Website